CLINICAL TRIAL: NCT02599051
Title: Transobturator Versus Single Incision Slings: 1 Year Results of a Randomized Control Trial
Brief Title: Transobturator Verus Single Incision Slings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cecilia Calvo (Other)
Responsible Party: Sponsor-Investigator, Cecilia Calvo, coordinator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 9034
Record Dates: First submitted 2015-11-03; First posted 2015-11-06 (Estimated); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monarc (Active Comparator): Placement of a transobturator monarc sling for stress urinary incontinence
  Interventions: Device: Monarc
- Mini-arc (Experimental): Placement of a single incision mini-arc sling for stress urinary incontinence
  Interventions: Device: Mini-arc

INTERVENTIONS:
Device: Mini-arc — We will place a single incision sling at the time of surgery for stress urinary incontinence
  Other Names: single incision sling
  Arms: Mini-arc
Device: Monarc — We will place a transobturator sling at the time of surgery for stress urinary incontinence
  Other Names: transobturator sling
  Arms: Monarc

SUMMARY:
A randomized control trial to compare the efficacy of the single incision mini-sling to the transobturator sling

DETAILED DESCRIPTION:
Transobturator slings are one type of sling that has become standard treatment for stress urinary incontinence. However, this procedure involves a total of 3 incisions to perform.

In contrast, single incision slings have been developed to treat stress urinary incontinence by using only one incision.

However, to date the success and complications of these two procedures have not been compared or studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urodynamically proven stress urinary incontinence who were planning on undergoing surgery for treatment.

Exclusion Criteria:

* Patients with prior incontinence surgery, a urodynamic diagnosis of intrinsic sphincter deficiency and mixed incontinence with a predominance of detrusor overactivity were excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G Willy Davila, MD, Principal Investigator — Cleveland Clinic Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Monarc | Mini-arc
Started | 49 | 49
Completed | 42 | 41
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monarc | Mini-arc | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 49 | 98
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 48.9 [39 to 57] | 52.9 [41 to 63] | 50 [39 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 49 | 98

OUTCOME MEASURES:

1. Primary Outcome: Objective Stress Urinary Incontinence
Description: The primary outcome was presence of leakage during cough stress test(CST) on examination
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Monarc | Mini-arc
Number analyzed (Participants) | 42 | 41
Participants | 9 | 12

2. Secondary Outcome: Quality of Life Questionnaire UDI-6
Description: Response to validated questionnaire: Urinary Distress Index(UDI-6) Measures symptoms on three subscales: 1. Irritative 2. Stress 3. Obstructive/Discomfort. The mean value of all questions answered is then multiplied by 25 for the actual score (range 0 to 100) Summary score - Add the scores from the 3 scales together to obtain the summary score (range 0 to 300) The higher the score the greater the perceived impact that pelvic floor dysfunction has on a patient's life.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monarc | Mini-arc
Number analyzed (Participants) | 42 | 41
score on a scale | 15.1 (16.4) | 20.3 (20.4)

3. Secondary Outcome: Subjective Patient Reported Recurrent or Persistent Stress Urinary Incontinence
Description: Assess if the patient has any complaint of stress urinary incontinence after surgery in follow up visits. This will be history only, no examination.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Monarc | Mini-arc
Number analyzed (Participants) | 42 | 41
participants | 11 | 21

4. Secondary Outcome: Number of Participants Who Completed Self- Assessment of Cure
Description: Self-assessment of cure is based on 5 point scale, cured, greatly improved, somewhat improved, not improved, and worsened. This is calculated by the number of patients that were analyzed.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Monarc | Mini-arc
Number analyzed (Participants) | 42 | 41
Participants | 37 | 31

5. Secondary Outcome: Quality of Life Questionnaire IIQ-7
Description: Response to validated questionnaire: Incontinence Impact Questionnaire(IIQ-7) The IIQ measures the impact of urinary incontinence on activities roles, and emotional states. A mean score is derived from each domain, then transferred to give weight to each subscale. Subscale scores range from 0-100. The total IIQ score is calculated by adding the four subscales score with a range of 0-400 possible. A score closer to 0 represents activities not affected at all versus closer to 400 represent activities that were greatly affected.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monarc | Mini-arc
Number analyzed (Participants) | 42 | 41
score on a scale | 8.95 (17.9) | 12.7 (20.8)

6. Secondary Outcome: Quality of Life Questionnaire ICIQ
Description: Response to validated questionnaire: International Consultation on Incontinence Questionnaire(ICIQ). The ICIQ is a screening tool for incontinence. The scoring scale is 0-21, minimum 0, maximum 21. a higher score indicates greater impairment from incontinence.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Monarc | Mini-arc
Number analyzed (Participants) | 42 | 41
scores on a scale | 3.1 (3.8) | 3.9 (4.3)

ADVERSE EVENTS:
Arm/Group | Monarc | Mini-arc
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 2/49 | 5/49
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monarc (N=49) | Mini-arc (N=49)
sling transectio (Surgical and medical procedures) | 1 (1) | 1 (1)
mesh exposure (Surgical and medical procedures) | 1 (1) | 3 (3)
dyspareunia (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No